CLINICAL TRIAL: NCT05188768
Title: Clinical Effects of Concentrated Growth Factor and Platelet-Rich Fibrin in the Treatment of Localized Gingival Recessions: A Split-Mouth Randomized Clinical Trial
Brief Title: Growth Factors in the Localized Gingival Recessions Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Seyma Bozkurt Doğan, Associate Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36290600/38
Record Dates: First submitted 2021-12-25; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Localized Gingival Recession
Keywords: localized gingival recession; Platelet rich fibrin; concentrated growth factor; coronally advanced flap

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentrated growth Factor Membrane (Experimental): Autogenous platelet and leukocyte fibrin material was obtained from blood.
  Interventions: Procedure: Concentrated Growth Factor Membrane; Procedure: Platelet Rich Fibrin
- Platelet Rich Fibrin (Active Comparator): Autogenous platelet and leukocyte fibrin material was obtained from blood.
  Interventions: Procedure: Concentrated Growth Factor Membrane; Procedure: Platelet Rich Fibrin

INTERVENTIONS:
Procedure: Concentrated Growth Factor Membrane — Concentrated growth factor is produced by the centrifugation of venous blood and platelets are concentrated in a gel layer containing fibrin matrix
  Other Names: An agent of platelet concentrates
Procedure: Platelet Rich Fibrin — Platelet Rich Fibrinis produced by the centrifugation of venous blood and platelets are concentrated in a gel layer containing fibrin matrix
  Other Names: An agent of platelet concentrates

SUMMARY:
The purpose of this study was to evaluate the clinical efficacy of concentrated-growth-factor (CGF) in combination with coronally-advanced-flap (CAF) compared with platelet-rich-fibrin (PRF)+CAF for the treatment of localized gingival-recessions (GRs)

DETAILED DESCRIPTION:
Gingival recession (GR) is a common mucogingival deformity. The root surface (RS) exposed by GR is treated with various surgical techniques.Traditionally, if GT and height of the keratinized gingiva (KG) are sufficient, the coronally advanced flap (CAF) technique is commonly used to close the exposed RS.Platelets contain various growth factors (GFs) to initiate healing process or regeneration of tissue.The second generation of platelet concentrates is platelet-rich fibrin (PRF) that are obtained from the centrifugation of blood (2700/3000rpm for 12 min) without anticoagulant or bovine trombin.And, the third generation of platelets concentrates is concentrated growth factor (CGF) as a new approach to produce PRF.It stated that the modified speed during centrifugation contribute the dense fibrin matrix in which includes larger, more intensive, more GFs than PRF.CGF is considered to be a biomaterial that is better than PRF in bone regeneration, but there is no study compare the clinical effects of CGF and PRF in the treatment of localized GRs. Our study hypothesized that if CGF has better regenerative capacity than PRF, the use of CGF in the treatment of GRs as a natural biomaterial may enhace the percentage of RC or healing of soft tissue compared with PRF. Therefore, the purpose of this study was to compare clinical effects of CGF and PRF in the treatment of localized GRs.

The patients of this randomized, split-mouth and controlled clinical trial study protocol were selected from individuals referred to the Department of Periodontology, at the Faculty of Dentistry, Bulent Ecevit University, for either dentin hypersensitivity or aesthetic complaints between April 2015 and June 2017.

The subjects were enrolled to this study based on the following inclusion criteria: (1) age > 18 years, (2) systemically and periodontally healthy, (3) non-smokers, (4) presence of ≥2 buccal adjacent Miller Class I or II GR with ≥2 mm GR depth (RD), probing depth (PD) <3 mm and gingival thickness (GT) ≥1 mm on both sides of the maxillary arch, (5) width of keratinized gingiva (KGW) ≥2 mm, (6) presence of identiﬁable cemento-enamel junction CEJ, (7) central, lateral canine and premolar teeth with GRs in the maxilla (8) full-mouth plaque control record (PCR) ≤20% (O'Leary et al. 1972) and gingival index (GI) scores = 0 (Loe, 1967) and presence of tooth vitality and absence of caries, restorations and furcation involvement in the treated area.

All the subjects received oral hygiene instructions and full-mouth scaling were performed 1 month before surgery. They were instructed to perform a non-traumatic brushing technique (Roll) using an ultra-soft toothbrush. In eighteen patients (mean age 39.67₊10.25 age; 8 females, 10 males), one side of the jaw received PRF+ CAF (37 defects), the opposite site received CGF + CAF (39 defects).

Application of PRF membrane to the control region: The patient's venous blood was taken into the 10-ml test tubes and placed quickly in the Electro-Mag centrifuge (M 815 P, İstanbul, Turkey) without shaking. The device was operated at 2700 rpm for 12 minutes to obtain PRF. Application of CGF membrane to the test region: The intravenous blood of the patient was taken into 10-ml glaas-coated test tubes without anticoagulant solutions and rapidly centrifuged with a CGF centrifuge machine (Medifuge, Silfradent, S. Sofia, Italy). The instrument's CGF program was selected and operated at speeds and angles ranging from 2700 to 3000 rpm. After approximately 13 minutes of rotation, CGF was obtained. CGF is characterized by 4 phases: (1) serum in the top layer, (2) the second buffy coat layer, (3) the third GF and unipotent stem cell layer (CGF), (4) the lower red blood cell layer (RBC). The CGFand PRF clot was removed from the tube and separated from the RBC by using microsurgical scissors. The CGF was squeezed in a special box that produces membranes at a constant thickness of 1 mm.All surgeries were performed by the same expert periodontist during a single surgical session Gingival recession sites were randomly determined as either test or control site by tossing a coin immediately before the surgical procedure.

Sutures were removed after 10 days and plaque control was maintained by CHX for additional 2 weeks. The patients started brush the tooth at the end of the 3rd week and they were again instructed in mechanical tooth cleaning of the treated tooth using an ultra soft toothbrush and roll technique. Oral hygiene instructions were provided at each postoperative visit.

ELIGIBILITY:
Inclusion Criteria:

* systemically and periodontally healthy,
* non-smokers
* presence of Miller Class I and II gingival recession with ≥ 2 mm gingival recession depth , probing depth <3 mm and gingival thickness (GT) ≥ 1 mm on both sides of the maxillary arch
* width of keratinized gingiva ≥ 2mm
* presence of identifiable cemento-enamel junction
* full-mouth plaque index (PI) < 20 % and gingival index (GI) scores =1,
* presence of tooth vitality and absence of caries, restorations and furcation involvement in the treated area,

Exclusion Criteria:

* - patients who had systemic problems that wound contraindicate for periodontal surgery, - usage of medications known to interfere with healing and to cause gingival enlargement - recession defects associated with demineralization, deep abrasion,
* previous surgery in the defects area within the past 1 year,
* pregnant or lactating females
* drug and alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Complete root coverage | 6 months
  Change from baseline in percentage of complete root coverage at 6th months.

SECONDARY OUTCOMES:
Percentage of mean root coverage | 6 months
  Change from baseline in percentage ofmean root coverage at 6th months.
Keratinized gingiva width | 6 months
  The distance is from the cemento-enamel junction to the gingival margin
Recession depth | 6 th months
  The distance is from the cemento-enamel junction to the gingival margin